CLINICAL TRIAL: NCT00133003
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of the Glycoprotein IIb/IIIa Inhibition With Abciximab in Patients With ACS Undergoing Coronary Stenting After Pretreatment With a High Loading Dose of Clopidogrel (ISAR-REACT-2)
Brief Title: Abciximab, Clopidogrel and Percutaneous Coronary Intervention in Acute Coronary Syndrome (ISAR-REACT-2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Deutsches Herzzentrum Muenchen, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A00500
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Disease; Angina, Unstable
MeSH Terms: conditions — Coronary Disease; Angina, Unstable | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Abciximab
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abciximab — 0.25 mg/kg of body weight bolus, followed by a 0.125-microg/kg per minute [maximum, 10 microg/min] infusion for 12 hours, plus heparin, 70 U/kg of body weight
  Other Names: ReoPro
  Arms: 1
Drug: Placebo — Placebo consist of placebo bolus and infusion of 12 hours (NaCl 0.9%), plus heparin bolus, 140 U/kg of body weight
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether there is any additional benefit from abciximab administration during percutaneous coronary intervention in patients presenting with acute coronary syndromes after pre-treatment with 600mg of clopidogrel.

DETAILED DESCRIPTION:
Although percutaneous coronary interventions (PCIs) are an established therapeutic approach in patients presenting with acute coronary syndrome (ACS), it is still unclear which the best antithrombotic therapy to be applied periprocedurally is. The EPISTENT trial has shown that adding abciximab (a glycoprotein [GP] IIb/IIIa receptor inhibitor) to the therapy with ticlopidine plus aspirin significantly reduces the incidence of ischemic complications (death, myocardial infarction or reinterventions) after coronary stent implantation. Ticlopidine also reduces procedural complications but has a delayed onset of action after coronary stenting and has been replaced by clopidogrel, which provides similar efficacy and is associated with fewer side effects. Experimental studies have shown that a 600 mg loading dose of clopidogrel is safe and acts rapidly leading to a maximal inhibition of platelet aggregation within 2 hours after administration. In the ISAR-REACT trial, a 600 mg loading dose of clopidogrel was well tolerated, and associated with such a low frequency of early complications that the use of abciximab offered no clinically measurable benefit at 30 days. Although patients with ACS have frequently been treated with a "cooling-off" strategy for >48 hours before undergoing PCI, the ISAR-COOL trial demonstrated that patients undergoing PCI within 6-12 hours of presentation with an ACS actually suffer a lower rate of ischemic complications than those for whom an invasive approach is delayed. However, patients with ACS represent a higher risk subset and may need a more potent antithrombotic regimen periprocedurally. Therefore, the results of ISAR REACT, which was performed in low and intermediate risk patients, should not be generalized to high risk patients.

Comparison:

All patients with non-ST-segment elevation acute coronary syndromes who will undergo coronary angiography willing to participate in the trial will receive a loading dose of 600 mg clopidogrel at least 2 hours prior to the procedure. Eligible patients who do not meet the exclusion criteria in whom angiography reveals that PCI is planned will be randomized to receive either abciximab plus low-dose heparin, 70 units/kg, or high dose heparin (140 units/kg) plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndromes
* Pretreatment (2 hours) with high loading dose (600 mg) clopidogrel
* Significant angiographic lesions amenable to and requiring a PCI
* Written informed consent

Exclusion Criteria:

* ST-segment elevation acute myocardial infarction within 48 hours from symptom onset
* Hemodynamic instability
* Pericarditis
* Malignancies with life expectancy less than one year
* Increased risk of bleeding
* Oral anticoagulation therapy with coumarin derivative within 7 days
* Recent use of GPIIb/IIIa inhibitors within 14 days
* Severe uncontrolled hypertension >180 mmHg unresponsive to therapy
* Relevant hematologic deviations: hemoglobin < 100g/L or hematocrit < 34%; platelet count < 100 x 10^9/L or platelet count > 600 x 10^9/L.
* Known allergy to the study medication
* Pregnancy (present or suspected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2022 (Actual)
Dates: Start 2003-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Composite rate of death, myocardial infarction, and urgent target vessel revascularization within 30 days | 30 days

SECONDARY OUTCOMES:
Major and minor bleeding complications in-hospital | in hospital
Death or myocardial infarction by 12 months | 12 months
Target vessel revascularization by 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Peter B Berger, MD, Study Director — Duke Clinical Research Institute
Locations (5):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Germany (3):
  - Herz-Zentrum, Bad Krozingen
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich
- St. Antonius Ziekenhuis Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Background] Topol EJ, Mark DB, Lincoff AM, Cohen E, Burton J, Kleiman N, Talley D, Sapp S, Booth J, Cabot CF, Anderson KM, Califf RM. Outcomes at 1 year and economic implications of platelet glycoprotein IIb/IIIa blockade in patients undergoing coronary stenting: results from a multicentre randomised trial. EPISTENT Investigators. Evaluation of Platelet IIb/IIIa Inhibitor for Stenting. Lancet. 1999 Dec 11;354(9195):2019-24. doi: 10.1016/s0140-6736(99)10018-7. PMID 10636365
- [Background] Topol EJ, Moliterno DJ, Herrmann HC, Powers ER, Grines CL, Cohen DJ, Cohen EA, Bertrand M, Neumann FJ, Stone GW, DiBattiste PM, Demopoulos L; TARGET Investigators. Do Tirofiban and ReoPro Give Similar Efficacy Trial. Comparison of two platelet glycoprotein IIb/IIIa inhibitors, tirofiban and abciximab, for the prevention of ischemic events with percutaneous coronary revascularization. N Engl J Med. 2001 Jun 21;344(25):1888-94. doi: 10.1056/NEJM200106213442502. PMID 11419425
- [Background] Neumann FJ, Kastrati A, Pogatsa-Murray G, Mehilli J, Bollwein H, Bestehorn HP, Schmitt C, Seyfarth M, Dirschinger J, Schomig A. Evaluation of prolonged antithrombotic pretreatment ("cooling-off" strategy) before intervention in patients with unstable coronary syndromes: a randomized controlled trial. JAMA. 2003 Sep 24;290(12):1593-9. doi: 10.1001/jama.290.12.1593. PMID 14506118
- [Background] Muller I, Seyfarth M, Rudiger S, Wolf B, Pogatsa-Murray G, Schomig A, Gawaz M. Effect of a high loading dose of clopidogrel on platelet function in patients undergoing coronary stent placement. Heart. 2001 Jan;85(1):92-3. doi: 10.1136/heart.85.1.92. No abstract available. PMID 11119474
- [Background] Pache J, Kastrati A, Mehilli J, Gawaz M, Neumann FJ, Seyfarth M, Hall D, Braun S, Dirschinger J, Schomig A. Clopidogrel therapy in patients undergoing coronary stenting: value of a high-loading-dose regimen. Catheter Cardiovasc Interv. 2002 Apr;55(4):436-41. doi: 10.1002/ccd.10092. PMID 11948888
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Result] Kastrati A, Mehilli J, Neumann FJ, Dotzer F, ten Berg J, Bollwein H, Graf I, Ibrahim M, Pache J, Seyfarth M, Schuhlen H, Dirschinger J, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic: Regimen Rapid Early Action for Coronary Treatment 2 (ISAR-REACT 2) Trial Investigators. Abciximab in patients with acute coronary syndromes undergoing percutaneous coronary intervention after clopidogrel pretreatment: the ISAR-REACT 2 randomized trial. JAMA. 2006 Apr 5;295(13):1531-8. doi: 10.1001/jama.295.13.joc60034. Epub 2006 Mar 13. PMID 16533938
- [Derived] Ndrepepa G, Kastrati A, Mehilli J, Neumann FJ, ten Berg J, Bruskina O, Dotzer F, Seyfarth M, Pache J, Dirschinger J, Ulm K, Berger PB, Schomig A. Age-dependent effect of abciximab in patients with acute coronary syndromes treated with percutaneous coronary interventions. Circulation. 2006 Nov 7;114(19):2040-6. doi: 10.1161/CIRCULATIONAHA.106.642306. Epub 2006 Oct 23. PMID 17060377